CLINICAL TRIAL: NCT03324698
Title: The Natural History of Chronic Pancreatitis: A Multicenter Study
Brief Title: The Natural History of Chronic Pancreatitis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Shenzhen People's Hospital (Other); Zhongda Hospital (Other); Qingdao University (Other); Jiangdu Hospital of Traditional Chinese Medicine (Unknown); Yangzhou University (Other); 307 Hospital of PLA (Other); The First People's Hospital of Hefei (Other); Nanjing PLA General Hospital (Other); The Second Artillery General Hospital (Other); Wulumuqi General Hospital of Lanzhou Military Command (Other); Central Hospital of Zaozhuang Mining Group (Unknown); Air Force General Hospital of the PLA (Other Government)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology Dept., Changhai Hospital
Other Study IDs: Changhai-171024
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Chronic Pancreatitis; Complication; Risk Factors
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic pancreatitis (CP) is a disease characterized by inflammation and their replacement by fibrotic tissue. The destruction of pancreatic function and structure are the main complications. This retrospective-prospective, multicenter, cohort study was conducted. This study aimed to observe the natural history of CP in China, analyse the risk factors for CP complications, and establish individual predictions.

DETAILED DESCRIPTION:
In order to track changes consistently throughout the course of CP and facilitate the evaluation and study of CP, a dedicated database, CP Database (version number 2.1, YINMA Information Technology Inc., Shanghai, China), was established to collect clinical data of CP patients who were admitted to our centers. Data befor CP Database established were retrospectively collected according to the electronic medical record system and complemented through telephone, letter, and e-mail inquiries. Data were prospectively collected since CP Database was established. The following information was documented in detail: demographic data (age, sex, birthplace, et al), course of CP, medical history, history of other diseases, smoking and alcohol history, family history of pancreatic diseases and diabetes mellitus (DM), laboratory and imaging findings, and treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic pancreatitis according to Asia-Pacific consensus

Exclusion Criteria:

* Pancreatic cancer diagnosed within 2 years after the diagnosis of chronic pancreatitis
* Groove pancreatitis
* Autoimmune pancreatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic pancreatitis patients in China
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2000-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Pancreatic cancer | Dec 31, 2017
  Pancreatic cancer developed in chronic pancreatitis patients
Diabetes mellitus | Dec 31, 2017
  Endocrine insufficiency developed in chronic pancreatitis patients
Steatorrhea | Dec 31, 2017
  Exocrine insufficiency developed in chronic pancreatitis patients
Pancreatic pseudocyst | Dec 31, 2017
  Pancreatic pseudocyst developed in chronic pancreatitis patients
Common bile duct stricture | Dec 31, 2017
  Common bile duct stricture developed in chronic pancreatitis patients

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Second Military Medical University, Shanghai, China

REFERENCES:
- [Background] Li BR, Pan J, Du TT, Liao Z, Ye B, Zou WB, Chen H, Ji JT, Zheng ZH, Wang D, Lin JH, Ning SB, Hu LH, Li ZS. Risk Factors for Steatorrhea in Chronic Pancreatitis: A Cohort of 2,153 Patients. Sci Rep. 2016 Feb 15;6:21381. doi: 10.1038/srep21381. PMID 26877248
- [Background] Hao L, Pan J, Wang D, Bi YW, Ji JT, Xin L, Liao Z, Du TT, Lin JH, Zhang D, Zeng XP, Ye B, Zou WB, Chen H, Xie T, Li BR, Zheng ZH, Hu LH, Li ZS. Risk factors and nomogram for pancreatic pseudocysts in chronic pancreatitis: A cohort of 1998 patients. J Gastroenterol Hepatol. 2017 Jul;32(7):1403-1411. doi: 10.1111/jgh.13748. PMID 28127800
- [Background] Hao L, Zeng XP, Xin L, Wang D, Pan J, Bi YW, Ji JT, Du TT, Lin JH, Zhang D, Ye B, Zou WB, Chen H, Xie T, Li BR, Zheng ZH, Wang T, Guo HL, Liao Z, Li ZS, Hu LH. Incidence of and risk factors for pancreatic cancer in chronic pancreatitis: A cohort of 1656 patients. Dig Liver Dis. 2017 Nov;49(11):1249-1256. doi: 10.1016/j.dld.2017.07.001. Epub 2017 Jul 15. PMID 28756974
- [Background] Hao L, Bi YW, Zhang D, Zeng XP, Xin L, Pan J, Wang D, Ji JT, Du TT, Lin JH, Ye B, Zou WB, Chen H, Xie T, Li BR, Zheng ZH, Wang T, Guo HL, Liao Z, Li ZS, Hu LH. Risk Factors and Nomogram for Common Bile Duct Stricture in Chronic Pancreatitis: A Cohort of 2153 Patients. J Clin Gastroenterol. 2019 Mar;53(3):e91-e100. doi: 10.1097/MCG.0000000000000930. PMID 28961573